CLINICAL TRIAL: NCT06533280
Title: A Multi-part Phase 1 Study Assessing the Safety, Tolerability, and PK of VH3739937 in Healthy Participants, by Conducting MAD and RBA Cohorts, With Optional Food Effect and Drug Interaction Cohorts
Brief Title: VH3739937 Phase 1 Multiple Ascending Dose (MAD) Study in Healthy Volunteers Including Relative Bioavailability (RBA), Optional Food Effect (FE), and Drug-drug Interaction (DDI)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 221773
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
Keywords: VH3739937; Multiple ascending dose; Relative bioavailability; Food effect; Drug-drug interaction
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind (sponsor-unblinded) study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part A MAD: VH3739937 (Experimental): Part A MAD: VH3739937 group will contain 3 ascending repeat-dose cohorts (Cohorts A1- A3), where participants will receive a twice daily (BID) dose of VH3739937 for 1 (Cohort A1), 2 (Cohort A2) or 3 (Cohort A3) days in fed conditions.
  Interventions: Drug: Part A, C and D: VH3739937 500 mg; Drug: Part A: VH3739937 100 mg
- Part A MAD: Placebo (Placebo Comparator): Part A MAD: Placebo group will include participants that will receive BID dose of placebo in fed conditions
  Interventions: Drug: Part A and C: Placebo
- Part B RBA/ optional FE: VH3739937 (Experimental): Part B RBA/FE: VH3739937 group will include participants that will receive treatment sequences (Treatment AB or BA) alternatively in Period 1 and Period 2 of the treatment. In Period 3 and Period 4, participants will receive 1 of 6 treatment sequences (CD, CE, ED, EC, DE, DC) in fed or fasted conditions.
  Interventions: Drug: Part B: Treatment A; Drug: Part B: Treatment B; Drug: Part B: Treatment C; Drug: Part B: Treatment D; Drug: Part B: Treatment E
- Part C: Optional QW VH3739937 (Experimental): Participants in this group will receive a weekly administration (QW) of VH3739937 during a 3-week period in fed conditions.
  Interventions: Drug: Part A, C and D: VH3739937 500 mg
- Part C: Optional QW Placebo (Placebo Comparator): Participants in this group will receive a weekly administration (QW) of placebo during a 3-week period in fed conditions.
  Interventions: Drug: Part A, C and D: VH3739937 500 mg; Drug: Part A and C: Placebo
- Part D: Optional DDI (Experimental): Participants in this group will receive a dose of the probe cocktail (Midazolam, Digoxin, Total Dabigatran etexilate, Rosuvastatin) alone on Day 1, followed by a subsequent dose of probe cocktail together with a single dose of VH3739937 on Day 10, in fed conditions.
  Interventions: Drug: Part A, C and D: VH3739937 500 mg; Drug: Part D: Probe cocktail

INTERVENTIONS:
Drug: Part A, C and D: VH3739937 500 mg — Oral administration of VH3739937 in moderate fat/moderate calorie conditions
  Arms: Part A MAD: VH3739937; Part C: Optional QW Placebo; Part C: Optional QW VH3739937; Part D: Optional DDI
Drug: Part A: VH3739937 100 mg — Oral administration of VH3739937 in moderate fat/moderate calorie conditions.
  Arms: Part A MAD: VH3739937
Drug: Part A and C: Placebo — Oral administration of Placebo in moderate fat/moderate calorie conditions
  Arms: Part A MAD: Placebo; Part C: Optional QW Placebo
Drug: Part B: Treatment A — VH3739937, 500 mg(single dose given as 5 x 100 mg tablets). administered under moderate fat/moderate calorie conditions (reference)
  Arms: Part B RBA/ optional FE: VH3739937
Drug: Part B: Treatment B — VH3739937, 500 mg (single dose given as 500 mg tablet) administered under moderate fat/moderate calorie conditions (test)
  Arms: Part B RBA/ optional FE: VH3739937
Drug: Part B: Treatment C — VH3739937, 500 mg single tablet administered under fasted conditions.
  Arms: Part B RBA/ optional FE: VH3739937
Drug: Part B: Treatment D — VH3739937, 500 mg single tablet administered under low-fat/ low calorie conditions.
  Arms: Part B RBA/ optional FE: VH3739937
Drug: Part B: Treatment E — VH3739937, 500 mg single tablet administered under high-fat/ high calorie conditions.
  Arms: Part B RBA/ optional FE: VH3739937
Drug: Part D: Probe cocktail — Oral administration of probe cocktail (Midazolam, Digoxin, Total Dabigatran etexilate, Rosuvastatin) in moderate fat/moderate calorie conditions.
  Arms: Part D: Optional DDI

SUMMARY:
This study will assess safety, tolerability and pharmacokinetic (PK) of VH3739937 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are overtly healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
2. Participants who can understand and comply with protocol requirements and timetables, instructions, and protocol-stated restrictions.

   Age
3. Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.

   Weight
4. Body weight >=50.0 kg (110 lbs) for men and >=45.0 kg (99 lbs) for women, and BMI within the range 18.5 to 32.0 kg/m2 (inclusive).

   Sex
5. Participants male at birth and participants female at birth:

   1. Participants male at birth:

      Participants male at birth are eligible to participate if they agree to the following during the study intervention period and for at least 90 days (a spermatogenesis cycle) after the last dose of study intervention:

      • Refrain from donating sperm

      PLUS either:

      • Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

      OR

      • Must agree to use contraception as detailed below: Agree to use a male condom and, if their partner is a person who is able to become pregnant, and who is not currently pregnant, they should also be advised of the benefit for their partner to use a highly effective method of contraception when having sexual intercourse, as a condom may break or leak.
   2. Participants female at birth:

   A participant who was female at birth is eligible to participate if they are not pregnant or breast- / chest- feeding, and one of the following conditions applies:

   • They are a PONCBP as defined in Section 10.4 Contraception and barrier guidance.

   The Investigator is responsible for review of medical history, menstrual history/postmenopausal status, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

   Informed consent
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

Exclusion Criteria:

Medical conditions

1. History or presence of cardiovascular, respiratory, hepatic, renal, GI, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
2. Unstable liver disease known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per Investigator assessment).
3. Known history of cirrhosis with or without viral hepatitis co-infection.
4. History of clinically relevant hepatitis within last 6 months.
5. Patients with chronic hepatitis B (HBsAg positive) infection (see HBV diagnostic criteria described below and in the study laboratory manual).
6. Have a history of malignant neoplasm (excepting definitively treated non-melanoma skin cancer or carcinoma in situ of the uterine cervix, which may be enrolled at any time) within the last 5 years.
7. Clinically significant cardiovascular disease.
8. A sustained semi-supine systolic blood pressure >150 mm Hg or <90 mm Hg or a semi-supine diastolic blood pressure >95 mm Hg or <50 mm Hg at Screening or Check-in.
9. A resting HR of <50 bpm or >100 bpm when vital signs are measured at Screening or Check-in. A HR from 100 bpm to 110 bpm can be rechecked by ECG or vital signs within up to 2 hours to verify eligibility.
10. An uninterpretable ECG or any significant arrhythmia or ECG finding which, in the opinion of the Investigator or VH/GSK Medical Monitor, will interfere with the safety of the individual participant.
11. Abnormalities on Screening ECG is allowed for eligibility determination: QTcF > 450 msec., QRS > 120 msec, PR > 220 msec
12. Any history of significant underlying psychiatric disorder, in the opinion of the Investigator or Medical Monitor; or a clinical assessment of suicidality based on the responses on the C-SSRS (Columbia Suicidality Scale). Participants' history of suicidal behaviour and/or suicidal ideation should be considered when evaluating for suicide risk.
13. Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the VH/GSK Medical Monitor.
14. Any pre-existing physical or other psychiatric condition which could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
15. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
16. A pre-existing condition, that could interfere with normal GI anatomy or motility hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study interventions or render the participant unable to take oral study intervention.

    Prior/Concomitant therapy
17. Past or intended use of over-the-counter or prescription medication within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing and for the duration of the study.
18. Use of narrow therapeutic index drugs that are substrates of P-gp or CYP3A are not permitted during the study.
19. Participants receiving any protocol-prohibited medication and who are unwilling or unable to switch to an alternate medication.

    Prior/Concurrent clinical study experience
20. Participation in the clinical study would result in loss of blood or blood products in excess of 500 mL within 56 days.
21. Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
22. Current enrollment or past participation in another investigational clinical study in which an investigational intervention was administered within the last either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent.
23. Past or current enrollment or past participation in earlier parts of this clinical study.

    Diagnostic assessments
24. Positive pre-enrollment clinical study drug/alcohol screen, including tetrahydrocannabinol.
25. Positive HIV fourth generation test.
26. Urine cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to Screening and at admission.
27. Any acute laboratory abnormality at Screening, which would preclude the participant's participation in the study of an investigational compound.
28. Any verified Grade 4 laboratory abnormality.
29. ALT >1.5 ULN or total bilirubin >1.5 ULN. Participants with Gilbert's syndrome can be included with total bilirubin >1.5xULN as long as direct bilirubin is <1.5xULN.
30. eGFR of <60 mL/min/1.73 m2 via CKD-EPI [Delgado, 2022].
31. Presence of HBsAg at Screening or within 3 months prior to first dose of study intervention.
32. Positive hepatitis C antibody test result at Screening or within 3 months prior to first dose of study intervention.
33. Positive hepatitis C RNA test result at Screening or within 3 months prior to first dose of study intervention.

    Other exclusion criteria
34. Regular alcohol consumption within 6 months prior to the clinical study.
35. Regular use of known drugs of abuse, including tetrahydrocannabinol.
36. Regular use of combustible tobacco products, and non-combustible nicotine delivery systems.
37. Sensitivity to heparin or heparin-induced thrombocytopenia.
38. Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that contraindicates participation in the clinical study.
39. Use of any products intended to treat medical conditions that are not approved by the governing health authority in a given country or region.
40. To assess any potential impact on participant eligibility with regard to safety, the Investigator must refer to the IB and supplements, approved product labels, and/or local prescribing information for detailed information regarding warnings, precautions, contraindications, AEs, drug interactions, and other significant data pertaining to the study drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with any adverse events (AEs) | Up to Day 25 for Cohorts A1 and A2 and Day 30 for Cohort A3
Part B: Number of participants with any adverse events (AEs) | Up to Day 15
Part C: Number of participants with any adverse events (AEs) | Up to Day 42
Part D: Number of participants with any adverse events (AEs) | Up to Day 28
Part A: Number of participants with adverse events (AEs) by grade of severity | Up to Day 25 for Cohorts A1 and A2, and Day 30 for Cohort A3
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part B: Number of participants with adverse events (AEs) by grade of severity | Up to Day 15 (Periods 2 and 4 only)
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part C: Number of participants with adverse events (AEs) by grade of severity | Up to Day 42
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part D: Number of participants with adverse events (AEs) by grade of severity | Up to Day 28
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part A: Number of participants with any serious adverse events (SAEs) | Up to Day 25 for Cohort A1 and A2 and Day 30 for Cohort A3
Part B: Number of participants with any serious adverse events (SAEs) | Up to Day 15 (Periods 2 and 4 only)
Part C: Number of participants with any serious adverse events (SAEs) | Up to Day 42
Part D: Number of participants with any serious adverse events (SAEs) | Up to Day 28
Part A: Number of participants with serious adverse events (SAEs) by grade of severity | Up to Day 25 for Cohort A1 and A2, and Day 30 for Cohort A3
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part B: Number of participants with serious adverse events (SAEs) by grade of severity | Up to Day 15 (Periods 2 and 4 only)
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part C: Number of participants with serious adverse events (SAEs) by grade of severity | Up to Day 42
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part D: Number of participants with serious adverse events (SAEs) by grade of severity | Up to Day 28
  The severity grade is defined as following: Grade 1= mild, Grade 2=moderate, Grade 3=severe, Grade 4=potentially life-threatening.
Part B: Area under the plasma concentration over a dosing interval from time of dosing to the time of the subsequent dose (AUC[0-t]) | At Days 1 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part B: AUC time curve from time zero to infinity (AUC[0-infinity]) | At Days 1 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part B: Time to maximum observed plasma concentration (Tmax) | At Days 1 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part B: Maximum observed plasma concentration (Cmax) after VH3739937 administration | At Days 1 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)

SECONDARY OUTCOMES:
Part B: AUC to the end of the dosing period (AUC[0-tau]) after VH3739937 administration | At Days 1, 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part B: AUC[0-infinity] after VH3739937 administration | At Days 1, 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part B: Tmax after VH3739937 administration | At Days 1, 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part B: Apparent terminal half-life (T1/2) after VH3739937 administration | At Days 1, 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part B: Apparent Oral Clearance (CL/F) after VH3739937 administration | At Days 1, 2, 3, 4, 6, 8, 12, 15 (Period 2 and Period 3 only)
Part D: AUC[0-tau] after VH3739937 administration | At Day 10 and Day 11
Part D: AUC[0-infinity] after VH3739937 administration | At Day 10 and Day 11
Part D: Cmax after VH3739937 administration | At Day 10 and Day 11
Part D: Tmax after VH3739937 administration | At Day 10 and Day 11
Part D: T1/2 after VH3739937 administration | At Day 10 and Day 11
Part D: CL/F after VH3739937 administration | At Day 10 and Day 11
Part A: AUC[0-tau] after VH3739937 administration | At Days 1 to 6, 8, 11, 15, 20, 25 (Cohort A1), at Days 1, 3 to 9, 11, 15, 20, 25 (Cohort A2), at Days 1, 4 to 8 , 10, 14, 18, 25, Day 30 (Cohort A3)
Part A: Cmax after VH3739937 administration | At Days 1 to 6, 8, 11, 15, 20, 25 (Cohort A1), at Days 1, 3 to 9, 11, 15, 20, 25 (Cohort A2), at Days 1, 4 to 8 , 10, 14, 18, 25, Day 30 (Cohort A3)
Part A: Tmax after VH3739937 administration | At Days 1 to 6, 8, 11, 15, 20, 25 (Cohort A1), at Days 1, 3 to 9, 11, 15, 20, 25 (Cohort A2), at Days 1, 4 to 8 , 10, 14, 18, 25, Day 30 (Cohort A3)
Part A: T1/2 after VH3739937 administration | At Days 1 to 6, 8, 11, 15, 20, 25 (Cohort A1), at Days 1, 3 to 9, 11, 15, 20, 25 (Cohort A2), at Days 1, 4 to 8 , 10, 14, 18, 25, Day 30 (Cohort A3)
Part C: AUC[0-tau] after VH3739937 administration | At Days 1, 2, 5, 7, 8, 9, 13, 15, 16, 17, 26, 34 and 42
Part C: Concentration in a dosing interval (Ctau) after VH3739937 administration | At Days 1, 2, 5, 7, 8, 9, 13, 15, 16, 17, 26, 34 and 42
Part C: Cmax after VH3739937 administration | At Days 1, 2, 5, 7, 8, 9, 13, 15, 16, 17, 26, 34 and 42
Part C: Tmax after VH3739937 administration | At Days 1, 2, 5, 7, 8, 9, 13, 15, 16, 17, 26, 34 and 42
Part C: T1/2 after VH3739937 administration | At Days 1, 2, 5, 7, 8, 9, 13, 15, 16, 17, 26, 34 and 42
Part C: CL/F after VH3739937 administration | At Days 1, 2, 5, 7, 8, 9, 13, 15, 16, 17, 26, 34 and 42
Part D: AUC[0-infinity] after probe cocktail administration | At Day 10 and Day 11
Part D: Cmax after probe cocktail administration | At Day 10 and Day 11
Part D: Tmax after probe cocktail administration | At Day 10 and Day 11
Part D: T1/2 after probe cocktail administration | At Day 10 and Day 11
Part D: CL/F after probe cocktail administration | At Day 10 and Day 11
Change from baseline for heart rate over all study groups | Up to Day 25 for Part A (Cohort A1 and A2) and Day 30 (Cohort A3), Day 15 for Part B, Day 17 and Day 42 for Part C, Day 14 and Day 28 for Part D
Change from baseline in PR Interval, QRS Interval, and QT Interval corrected for heart rate using Fridericias formula (QTcF) over all study groups | At Days (D) 1 to 5, 8, 15, 25 for Cohort A1 (Part A), D 1 to 6, 9, 15, 25 for Cohort A2 (Part A), D 1 to 7, 10, 18, 30 for Cohort A3 (Part A), at D 1, 3, 6, 12,15 for Part B, at D 1, 2, 8, 9, 13 to 17, 42 for Part C, at D 1, 3, 10, 14, 28 for Part D
Placebo-corrected change from baseline heart rate over alll study groups | At Days (D) 1 to 5, 8, 15, 25 for Cohort A1 (Part A), D 1 to 6, 9, 15, 25 for Cohort A2 (Part A), D 1 to 7, 10, 18, 30 for Cohort A3 (Part A), at D 1, 3, 6, 12,15 for Part B, at D 1, 2, 8, 9, 13 to 17, 42 for Part C, at D 1, 3, 10, 14, 28 for Part D
Placebo-corrected change from baseline in PR Interval, QRS Interval, and QT Interval corrected for heart rate using Fridericias formula (QTcF) over all study groups | At Days (D) 1 to 5, 8, 15, 25 for Cohort A1 (Part A), D 1 to 6, 9, 15, 25 for Cohort A2 (Part A), D 1 to 7, 10, 18, 30 for Cohort A3 (Part A), at D 1, 3, 6, 12,15 for Part B, at D 1, 2, 8, 9, 13 to 17, 42 for Part C, at D 1, 3, 10, 14, 28 for Part D
Categorical outliers for heart rate, PR Interval, QRS Interval and QT Interval over all study groups | At Days (D) 1 to 5, 8, 15, 25 for Cohort A1 (Part A), D 1 to 6, 9, 15, 25 for Cohort A2 (Part A), D 1 to 7, 10, 18, 30 for Cohort A3 (Part A), at D 1, 3, 6, 12,15 for Part B, at D 1, 2, 8, 9, 13 to 17, 42 for Part C, at D 1, 3, 10, 14, 28 for Part D
Frequency of treatment-emergent electrocardiogram (ECG) morphology changes over all study groups | At Days (D) 1 to 5, 8, 15, 25 for Cohort A1 (Part A), D 1 to 6, 9, 15, 25 for Cohort A2 (Part A), D 1 to 7, 10, 18, 30 for Cohort A3 (Part A), at D 1, 3, 6, 12,15 for Part B, at D 1, 2, 8, 9, 13 to 17, 42 for Part C, at D 1, 3, 10, 14, 28 for Part D

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/